CLINICAL TRIAL: NCT02760264
Title: A Phase IIa Open-Label, Multiple Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Exploratory Efficacy of Vamorolone in Boys With Duchenne Muscular Dystrophy (DMD)
Brief Title: A Study to Assess Vamorolone in Boys With Duchenne Muscular Dystrophy (DMD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ReveraGen BioPharma, Inc. (Industry)
Collaborators: University of Pittsburgh (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Cooperative International Neuromuscular Research Group (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VBP15-002; 1R44NS095423-01 (NIH); 1U34AR068616-01 (NIH)
Record Dates: First submitted 2016-04-28; First posted 2016-05-03 (Estimated); Results first posted 2019-01-02 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; vamorolone
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — VBP15 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dose Level Group 1 (Experimental): Participants enrolled in Dose Level Group 1 will receive vamorolone 0.25 mg/kg/day.
  Interventions: Drug: Vamorolone 0.25 mg/kg/day
- Dose Level Group 2 (Experimental): Participants enrolled in Dose Level Group 2 will receive vamorolone 0.75 mg/kg/day.
  Interventions: Drug: Vamorolone 0.75 mg/kg/day
- Dose Level Group 3 (Experimental): Participants enrolled in Dose Level Group 3 will receive vamorolone 2.0 mg/kg/day.
  Interventions: Drug: Vamorolone 2.0 mg/kg/day
- Dose Level Group 4 (Experimental): Participants enrolled in Dose Level Group 4 will receive vamorolone 6.0 mg/kg/day.
  Interventions: Drug: Vamorolone 6.0 mg/kg/day

INTERVENTIONS:
Drug: Vamorolone 0.25 mg/kg/day — Oral administration of 0.25 mg/kg/day daily for 14 days.
  Other Names: VBP15
  Arms: Dose Level Group 1
Drug: Vamorolone 0.75 mg/kg/day — Oral administration of 0.75 mg/kg/day daily for 14 days.
  Other Names: VBP15
  Arms: Dose Level Group 2
Drug: Vamorolone 2.0 mg/kg/day — Oral administration of 2.0 mg/kg/day daily for 14 days.
  Other Names: VBP15
  Arms: Dose Level Group 3
Drug: Vamorolone 6.0 mg/kg/day — Oral administration of 6 mg/kg/day daily for 14 days.
  Other Names: VBP15
  Arms: Dose Level Group 4

SUMMARY:
The purpose of this study is to determine whether a new medication called vamorolone is safe and well-tolerated by boys with Duchenne muscular dystrophy (DMD) ages ≥ 4 and < 7 years old.

DETAILED DESCRIPTION:
This study will evaluate the safety and tolerability of a new steroid-like medication called vamorolone in boys with DMD ages ≥ 4 years and < 7 years. Enrolled participants will take the study medication for 14 days followed by a 14 day follow-up period. The potential effectiveness of vamorolone in treating DMD will also be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's parent or legal guardian has provided written informed consent/Health Insurance Portability and Accountability Act (HIPAA) authorization prior to any study-related procedures;
2. Subject has a confirmed (by Central Genetic Counselor) diagnosis of DMD as defined as:

   1. Dystrophin immunofluorescence and/or immunoblot showing complete dystrophin deficiency, and clinical picture consistent with typical DMD, OR
   2. Identifiable mutation within the DMD gene (deletion/duplication of one or more exons) where reading frame can be predicted as 'out-of-frame', and clinical picture consistent with typical DMD, OR
   3. Complete dystrophin gene sequencing showing an alteration (point mutation, duplication, other) that is expected to preclude production of the dystrophin protein (i.e. nonsense mutation, deletion/duplication leading to a downstream stop codon), with a typical clinical picture of DMD;
3. Subject is ≥ 4 years and < 7 years of age at time of enrollment in the study;
4. Subject is able to complete the Time to Stand Test (TTSTAND) without assistance, as assessed at the Screening and Baseline Visits;
5. Clinical laboratory test results are within the normal range at the Screening Visit, or if abnormal, are not clinically significant, in the opinion of the Investigator. (Note: Serum gamma glutamyl transferase [GGT], creatinine, and total bilirubin all must be ≤ upper limit of the normal range at the Screening Visit);
6. Subject has evidence of chicken pox immunity as determined by presence of IgG antibodies to varicella, as documented by a positive test result from the testing laboratory at the Screening Visit; and
7. Subject and parent/guardian are willing and able to comply with scheduled visits, study drug administration plan, and study procedures.

Exclusion Criteria:

1. Subject has current or history of major renal or hepatic impairment, diabetes mellitus or immunosuppression;
2. Subject has current or history of chronic systemic fungal or viral infections;
3. Subject has had an acute illness within 4 weeks prior to the first dose of study medication;
4. Subject has used mineralocorticoid receptor agents, such as spironolactone, eplerenone, canrenone (canrenoate potassium), prorenone (prorenoate potassium), mexrenone (mexrenoate potassium) within 4 weeks prior to the first dose of study medication;
5. Subject has evidence of symptomatic cardiomyopathy. [Note: Asymptomatic cardiac abnormality on investigation would not be exclusionary];
6. Subject is currently being treated or has received previous treatment with oral glucocorticoids or other immunosuppressive agents. [Notes: Past transient use of oral glucocorticoids or other oral immunosuppressive agents for no longer than 3 months cumulative, with last use at least 3 months prior to first dose of study medication, will be considered for eligibility on a case-by-case basis. Inhaled and/or topical corticosteroids prescribed for an indication other than DMD are permitted but must be administered at stable dose for at least 3 months prior to study drug administration];
7. Subject has used idebenone within 4 weeks prior to the first dose of study medication;
8. Subject has an allergy or hypersensitivity to the study medication or to any of its constituents;
9. Subject has severe behavioral or cognitive problems that preclude participation in the study, in the opinion of the Investigator;
10. Subject has previous or ongoing medical condition, medical history, physical findings or laboratory abnormalities that could affect safety, make it unlikely that treatment and follow-up will be correctly completed or impair the assessment of study results, in the opinion of the Investigator;
11. Subject is taking any other investigational drug currently or has taken any other investigational drug within 3 months prior to the start of study treatment; or
12. Subject has previously been enrolled in the study.

Ages: 4 Years to 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 48 (Actual)
Dates: Start 2016-06; Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula R Clemens, MD, Study Chair — University of Pittsburgh
Locations (12):
- United States (6):
  - University of California Davis, Davis, California
  - University of Florida, Gainesville, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Ann & Robert H. Lurie Children's Hospital, Chicago, Illinois
  - Duke University, Durham, North Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Australia (2):
  - Royal Children's Hospital, Melbourne
  - Sydney Children's Hospital, Westmead
- Alberta Children's Hospital, Calgary, Alberta, Canada
- Schneider Children's Medical Center, Petah Tikvah, Israel
- Queen Silvia Children's Hospital, Gothenburg, Sweden
- Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hoffman E, Gaglianone S, Ketema R, Tu W, Peay H, Clemens P, Dang U, Conklin L. Return of participant-level clinical trial results to participants: pilot of a simplified centralised approach. BMJ Open. 2024 Mar 23;14(3):e080097. doi: 10.1136/bmjopen-2023-080097. PMID 38521535
- [Derived] Smith EC, Conklin LS, Hoffman EP, Clemens PR, Mah JK, Finkel RS, Guglieri M, Tulinius M, Nevo Y, Ryan MM, Webster R, Castro D, Kuntz NL, Kerchner L, Morgenroth LP, Arrieta A, Shimony M, Jaros M, Shale P, Gordish-Dressman H, Hagerty L, Dang UJ, Damsker JM, Schwartz BD, Mengle-Gaw LJ, McDonald CM; CINRG VBP15 and DNHS Investigators. Efficacy and safety of vamorolone in Duchenne muscular dystrophy: An 18-month interim analysis of a non-randomized open-label extension study. PLoS Med. 2020 Sep 21;17(9):e1003222. doi: 10.1371/journal.pmed.1003222. eCollection 2020 Sep. PMID 32956407
- [Derived] Li X, Conklin LS, van den Anker J, Hoffman EP, Clemens PR, Jusko WJ. Exposure-Response Analysis of Vamorolone (VBP15) in Boys With Duchenne Muscular Dystrophy. J Clin Pharmacol. 2020 Oct;60(10):1385-1396. doi: 10.1002/jcph.1632. Epub 2020 May 20. PMID 32434278
- See also: Cooperative International Research Group — http://cinrgresearch.org/
- See also: ReveraGen BioPharma, Inc — http://www.reveragen.com/
- See also: Phase IIa trial in Duchenne muscular dystrophy shows vamorolone is a first-in-class dissociative steroidal anti-inflammatory drug. — https://www.ncbi.nlm.nih.gov/pubmed/30219580

RESULTS

PARTICIPANT FLOW:
Groups:
- Vamorolone 0.25 mg/kg/Day: Participants enrolled in Dose Level Group 1 will receive vamorolone 0.25 mg/kg/day.
  Oral administration of 0.25 mg/kg/day daily for 14 days.
- Vamorolone 0.75 mg/kg/Day: Participants enrolled in Dose Level Group 2 will receive vamorolone 0.75 mg/kg/day.
  Oral administration of 0.75 mg/kg/day daily for 14 days.
- Vamorolone 2.0 mg/kg/Day: Participants enrolled in Dose Level Group 3 will receive vamorolone 2.0 mg/kg/day.
  Oral administration of 2.0 mg/kg/day daily for 14 days.
- Vamorolone 6.0 mg/kg/Day: Participants enrolled in Dose Level Group 4 will receive vamorolone 6.0 mg/kg/day.
  Oral administration of 6 mg/kg/day daily for 14 days.
Period: 0.25 mg/kg/Day
Arm/Group | Vamorolone 0.25 mg/kg/Day | Vamorolone 0.75 mg/kg/Day | Vamorolone 2.0 mg/kg/Day | Vamorolone 6.0 mg/kg/Day
Started | 12 | 0 | 0 | 0
Completed | 12 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: 0.75 mg/kg/Day
Arm/Group | Vamorolone 0.25 mg/kg/Day | Vamorolone 0.75 mg/kg/Day | Vamorolone 2.0 mg/kg/Day | Vamorolone 6.0 mg/kg/Day
Started | 0 | 12 | 0 | 0
Completed | 0 | 12 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: 2.0 mg/kg/Day
Arm/Group | Vamorolone 0.25 mg/kg/Day | Vamorolone 0.75 mg/kg/Day | Vamorolone 2.0 mg/kg/Day | Vamorolone 6.0 mg/kg/Day
Started | 0 | 0 | 12 | 0
Completed | 0 | 0 | 12 | 0
Not Completed | 0 | 0 | 0 | 0
Period: 6.0 mg/kg/Day
Arm/Group | Vamorolone 0.25 mg/kg/Day | Vamorolone 0.75 mg/kg/Day | Vamorolone 2.0 mg/kg/Day | Vamorolone 6.0 mg/kg/Day
Started | 0 | 0 | 0 | 12
Completed | 0 | 0 | 0 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4 | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 48
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 5.2 (1.03) | 4.8 (0.83) | 4.7 (0.89) | 4.8 (0.75) | 4.9 (0.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 12 | 12 | 12 | 12 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 3 | 4
  Not Hispanic or Latino | 12 | 11 | 12 | 9 | 44
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 11 | 10 | 12 | 12 | 45
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 3 | 0 | 2 | 2 | 7
  Sweden | 0 | 4 | 0 | 0 | 4
  United States | 9 | 3 | 2 | 6 | 20
  United Kingdom | 0 | 0 | 4 | 2 | 6
  Israel | 0 | 3 | 2 | 0 | 5
  Australia | 0 | 2 | 2 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Summary of Adverse Events as Assessed by CTCAE Version 4.03
Description: Treatment-emergent adverse events (TEAEs) are defined as any adverse event or worsening of an existing conditions after initiation of the investigational product and through the subject's last study visit (study completion or early termination). Serious adverse events were recorded for up to 30 days after the final administration of study drug.
  Note: Total Number of Treatment Emergent Adverse Events: The total incidences of TEAEs experienced in study; Any Treatment Emergent Adverse Event: TEAEs reported at least once per dose group
Time Frame: Adverse events will be recorded from the date of informed consent and through the time of the subject's last study visit. Serious adverse events will be recorded from the date of informed consent and for up to 30 days after final drug administration.
Population: Safety Population: All subjects who receive at least one dose of vamorolone study medication will be included in safety population.
Measure: Number; unit: Number of Events
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 12 | 12 | 12 | 12
Number of Events
  Total Number of Adverse Events | 16 | 18 | 13 | 11
  Total Number of Treatment Emergent Adverse Events | 13 | 13 | 11 | 9
  Any Treatment Emergent Adverse Events | 7 | 6 | 8 | 7
  Any Drug Related Treatment Emergent Adverse Events | 1 | 2 | 2 | 3
  Any CTCAE Grade 3 or Higher TEAE | 0 | 0 | 0 | 0
  Discontinuation of Study Drug due to TEAE | 0 | 0 | 0 | 0
  Any Serious Treatment Emergent Adverse Events | 0 | 0 | 0 | 0
  Death | 0 | 0 | 0 | 0

2. Secondary Outcome: Serum Pharmacodynamic Biomarkers (Insulin Resistance)- Fasting Glucose
Description: Pharmacodynamic biomarkers were measured to investigate the effects of single and multiple oral doses of vamorolone on serum PD biomarkers in ambulant boys ages 4-< 7 years with DMD.
Time Frame: Baseline, Week 2
Population: Safety Population: All subject who receive at least dose of vamorolone study medication will be included in the safety population.
Measure: Mean (Standard Deviation); unit: mg/ dL
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 12 | 12 | 12 | 12
mg/ dL
  Baseline: number analyzed (Participants) | 12 | 12 | 12 | 10
  Baseline | 87.5 (9.44) | 88.9 (18.71) | 89.3 (7.91) | 92.3 (8.19)
  Week 2 | 85.3 (9.29) | 83.1 (6.69) | 89.5 (5.20) | 89.2 (11.12)
  Week 2 Change from Baseline: number analyzed (Participants) | 12 | 12 | 12 | 10
  Week 2 Change from Baseline | -2.2 (10.46) | -5.8 (18.92) | 0.2 (8.79) | -1.3 (9.41)
Statistical Analysis 1: Comparison: Dose Level Group 1 vs Dose Level Group 2 vs Dose Level Group 3 vs Dose Level Group 4; Test type: Other — Treatment levels were not compared; Safety Population was used for this analysis. Safety Population includes all subjects who receive at least one dose of vamorolone study medication. Treatment levels were not compared

3. Secondary Outcome: Serum Pharmacodynamic Biomarkers (Insulin Resistance) -Fasting Glucose
Description: as for outcome 2
Time Frame: Baseline, Week 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Week 2 % change from Baseline
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 12 | 12 | 12 | 10
Week 2 % change from Baseline | -1.8 (13.07) | -4.2 (13.98) | 0.8 (9.76) | -1.2 (9.80)

4. Secondary Outcome: Serum Pharmacodynamic Biomarkers (Insulin Resistance)- Insulin
Description: as for outcome 2
Time Frame: Baseline , Week 2
Population: Safety Population All subjects who receive at least one dose of vamorolone study medication will be included in the Safety Population.
Measure: Mean (Standard Deviation); unit: µIU/mL
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 12 | 12 | 12 | 12
µIU/mL
  Baseline: number analyzed (Participants) | 11 | 8 | 12 | 12
  Baseline | 5.54 (3.651) | 3.09 (2.033) | 3.40 (1.548) | 3.96 (2.027)
  Week 2: number analyzed (Participants) | 11 | 11 | 12 | 12
  Week 2 | 5.29 (2.671) | 3.22 (1.924) | 3.87 (2.118) | 6.73 (4.599)
  Week 2 Change from Baseline: number analyzed (Participants) | 10 | 8 | 12 | 12
  Week 2 Change from Baseline | -0.65 (2.913) | 0.34 (1.289) | 0.47 (2.777) | 2.78 (4.651)
Statistical Analysis 1: Comparison: Dose Level Group 1 vs Dose Level Group 2 vs Dose Level Group 3 vs Dose Level Group 4; Test type: Other — Treatment levels were not compared; [other analysis details as in outcome 2, analysis 1]

5. Secondary Outcome: Serum Pharmacodynamic Biomarkers (Insulin Resistance)- Insulin
Description: as for outcome 2
Time Frame: Baseline, Week 2
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Week 2 % change from Baseline
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 10 | 8 | 12 | 12
Week 2 % change from Baseline | -5.54 (32.622) | 26.07 (76.483) | 42.85 (107.337) | 83.55 (117.064)

6. Secondary Outcome: Serum Pharmacodynamic Biomarkers (Adrenal Axis Suppression)- First in Morning Cortisol
Description: as for outcome 2
Time Frame: Week 2 (pre-dose)
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 11 | 11 | 11 | 10
mcg/dL | 10.425 (1.7358) | 9.755 (2.7614) | 7.321 (3.0322) | 3.010 (1.0141)
Statistical Analysis 1: Comparison: Dose Level Group 1 vs Dose Level Group 2 vs Dose Level Group 3 vs Dose Level Group 4; Test type: Other — Treatment levels were not compared; [other analysis details as in outcome 2, analysis 1]

7. Secondary Outcome: Serum Pharmacodynamics Biomarkers (Bone Turnover) -Osteocalcin
Description: as for outcome 2
Time Frame: Baseline, Day 1, Week 2, Week 4
Population: Safety Population: All subjects who receive at least one dose of vamorolone study medication will be included in the Safety Population.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 12 | 12 | 12 | 12
ng/mL
  Baseline | 37.94 (11.622) | 35.66 (6.800) | 41.17 (5.617) | 44.36 (5.979)
  Day 1: number analyzed (Participants) | 12 | 12 | 12 | 11
  Day 1 | 39.37 (14.189) | 35.89 (7.526) | 34.93 (6.881) | 33.52 (9.135)
  Day 1 Change from Baseline: number analyzed (Participants) | 12 | 12 | 12 | 11
  Day 1 Change from Baseline | 1.43 (8.197) | 0.23 (5.304) | -6.23 (10.930) | -11.37 (9.137)
  Week 2 | 38.53 (12.025) | 35.10 (8.238) | 37.51 (8.624) | 29.04 (4.853)
  Week 2 Change from Baseline | 0.58 (5.986) | -0.56 (7.934) | -3.66 (9.818) | -15.32 (6.450)
  Week 4 | 39.20 (14.136) | 42.24 (8.426) | 47.91 (6.648) | 42.81 (10.851)
  Week 4 Change from Baseline | 1.26 (5.650) | 6.58 (9.341) | 6.74 (9.747) | -1.55 (11.176)
Statistical Analysis 1: Comparison: Dose Level Group 1 vs Dose Level Group 2 vs Dose Level Group 3 vs Dose Level Group 4; Test type: Other — Treatment levels were not compared; [other analysis details as in outcome 2, analysis 1]

8. Secondary Outcome: Serum Pharmacodynamics Biomarkers (Bone Turnover) -Osteocalcin
Description: as for outcome 2
Time Frame: Baseline, Day 1, Week 2, Week 4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: % change from Baseline
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 12 | 12 | 12 | 12
% change from Baseline
  Day 1 Percent Change from Baseline: number analyzed (Participants) | 12 | 12 | 12 | 11
  Day 1 Percent Change from Baseline | 3.95 (22.015) | 1.41 (15.449) | -12.63 (25.020) | -25.05 (20.228)
  Week 2 Percent Change from Baseline | 2.48 (16.756) | -0.07 (22.408) | -7.81 (23.664) | -33.87 (12.548)
  Week 4 Percent Change from Baseline | 2.72 (14.063) | 20.91 (28.644) | 18.74 (25.095) | -2.43 (25.932)

9. Secondary Outcome: Serum Pharmacodynamic Biomarkers (Bone Turnover)- Procollagen 1 N-Terminal Propeptide
Description: as for outcome 2
Time Frame: Baseline Day 1 Week 2 Week 4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 12 | 12 | 12 | 12
ng/mL
  Baseline: number analyzed (Participants) | 12 | 11 | 12 | 12
  Baseline | 555.8 (184.72) | 480.7 (118.20) | 508.2 (94.36) | 511.5 (106.50)
  Day 1: number analyzed (Participants) | 12 | 12 | 12 | 11
  Day 1 | 474.0 (116.45) | 443.7 (112.38) | 417.1 (87.35) | 475.2 (147.10)
  Day 1 Change from Baseline: number analyzed (Participants) | 12 | 11 | 12 | 11
  Day 1 Change from Baseline | -81.8 (124.24) | -34.5 (101.97) | -91.1 (64.64) | -36.5 (144.04)
  Week 2 | 443.8 (93.86) | 407.8 (96.54) | 346.6 (68.59) | 303.7 (56.38)
  Week 2 Change from Baseline: number analyzed (Participants) | 12 | 11 | 12 | 12
  Week 2 Change from Baseline | -112.0 (125.08) | -70.6 (123.69) | -161.6 (73.52) | -207.8 (78.16)
  Week 4 | 573.8 (251.02) | 496.7 (117.57) | 492.0 (81.92) | 566.3 (149.32)
  Week 4 Change from Baseline: number analyzed (Participants) | 12 | 11 | 12 | 12
  Week 4 Change from Baseline | 18.1 (153.10) | 21.3 (122.87) | -16.2 (79.64) | 54.8 (118.09)
Statistical Analysis 1: Comparison: Dose Level Group 1 vs Dose Level Group 2 vs Dose Level Group 3 vs Dose Level Group 4; Test type: Other — Treatment levels were not compared; [other analysis details as in outcome 2, analysis 1]

10. Secondary Outcome: Serum Pharmacodynamic Biomarkers (Bone Turnover)- Procollagen 1 N-Terminal Propeptide
Description: as for outcome 2
Time Frame: Baseline, Day 1, Week 2, Week 4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: % change from Baseline
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 12 | 12 | 12 | 12
% change from Baseline
  Day 1 Percent Change from Baseline: number analyzed (Participants) | 12 | 11 | 12 | 11
  Day 1 Percent Change from Baseline | -12.2 (17.07) | -5.4 (24.58) | -17.4 (12.59) | -5.7 (30.76)
  Week 2 Percent Change from Baseline | -17.5 (14.65) | -11.2 (29.19) | -30.9 (11.80) | -39.9 (9.22)
  Week 4 Percent Change from Baseline | 2.8 (25.57) | 7.8 (30.86) | -1.4 (17.47) | 11.8 (28.24)

11. Secondary Outcome: Serum Pharmacodynamic Biomarkers (Bone Turnover)-Type I Collagen C-Telopeptides
Description: as for outcome 2
Time Frame: Baseline, Day 1, Week 4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 12 | 12 | 12 | 12
pg/mL
  Baseline: number analyzed (Participants) | 11 | 12 | 12 | 12
  Baseline | 871.0 (160.85) | 935.8 (286.50) | 936.8 (256.25) | 889.3 (186.68)
  Day 1: number analyzed (Participants) | 12 | 12 | 12 | 11
  Day 1 | 974.8 (252.77) | 940.8 (227.60) | 838.3 (233.30) | 786.8 (331.68)
  Day 1 Change from Baseline: number analyzed (Participants) | 11 | 10 | 12 | 11
  Day 1 Change from Baseline | 72.4 (241.87) | -12.9 (233.44) | -98.5 (237.69) | -115.7 (421.04)
  Week 2 | 963.7 (157.68) | 903.3 (251.01) | 710.4 (180.03) | 625.7 (203.19)
  Week 2 Change from Baseline: number analyzed (Participants) | 11 | 10 | 12 | 12
  Week 2 Change from Baseline | 85.0 (185.90) | -19.9 (266.99) | -226.4 (185.99) | -263.7 (229.69)
  Week 4 | 915.9 (263.13) | 983.5 (298.47) | 949.8 (303.76) | 989.2 (216.29)
  Week 4 Change from Baseline: number analyzed (Participants) | 11 | 10 | 12 | 12
  Week 4 Change from Baseline | 17.4 (267.45) | 34.8 (271.50) | 12.9 (181.45) | 99.8 (211.90)
Statistical Analysis 1: Comparison: Dose Level Group 1 vs Dose Level Group 2 vs Dose Level Group 3 vs Dose Level Group 4; Test type: Other — Treatment levels were not compared; [other analysis details as in outcome 2, analysis 1]

12. Secondary Outcome: Serum Pharmacodynamic Biomarkers (Bone Turnover)-Type I Collagen C-Telopeptides
Description: as for outcome 2
Time Frame: Baseline, Day 1, Week 4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: % change from Baseline
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 12 | 12 | 12 | 12
% change from Baseline
  Day 1 Percent Change from Baseline: number analyzed (Participants) | 11 | 10 | 12 | 11
  Day 1 Percent Change from Baseline | 9.9 (25.38) | 2.7 (23.76) | -8.0 (23.93) | -6.7 (53.72)
  Week 2 Percent Change from Baseline: number analyzed (Participants) | 11 | 10 | 12 | 12
  Week 2 Percent Change from Baseline | 11.9 (20.52) | 2.2 (26.44) | -22.5 (15.27) | -27.7 (26.50)
  Week 4 Percent Change from Baseline: number analyzed (Participants) | 11 | 10 | 12 | 12
  Week 4 Percent Change from Baseline | 3.6 (28.96) | 6.8 (24.06) | 2.7 (19.03) | 14.5 (32.98)

13. Secondary Outcome: Pharmacokinetic (PK) Assessments (Tmax)
Description: Plasma concentrations of vamorolone were measured using a specific and validated liquid chromatography tandem mass spectrometry (LC-MS) assay. tmax= time when plasma concentration is at maximum.
Time Frame: Day 1, Week 2
Population: All subjects who receive at least one dose of vamorolone study medication and have sufficient quantifiable plasma concentration data for PK analysis will be included in the PK population. [Note that the PK population will be determined by the study pharmacokineticist upon review of the concentration information for each subject in each cohort.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 11 | 12 | 12 | 12
hour
  Day 1 | 3.6 (1.2) | 4.6 (2.1) | 2.5 (1.3) | 2.7 (1.3)
  Week 2 | 3.8 (1.80) | 3.8 (2.2) | 2.8 (1) | 2.3 (0.86)

14. Secondary Outcome: Pharmacokinetic (PK) Assessments (AUC Inf)
Description: Plasma concentrations of vamorolone were measured using a specific and validated liquid chromatography tandem mass spectrometry (LC-MS) assay. AUC inf= Area under the concentration vs. time curve to time infinity.
Time Frame: Day 1, Week 2
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: [(hr)(ng)/mL]
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 11 | 12 | 12 | 12
[(hr)(ng)/mL]
  Day 1 | 118 (48) | 379 (117) | 761 (352) | 3279 (1693)
  Week 2 | 164 (61) | 544 (155) | 1138 (467) | 3606 (897)

15. Secondary Outcome: Pharmacokinetic (PK) Assessments CL (ml/hr/kg)
Description: Plasma concentrations of vamorolone were measured using a specific and validated liquid chromatography tandem mass spectrometry (LC-MS) assay
Time Frame: Day 1, Week 2
Measure: Mean (Standard Deviation); unit: ml/hr/kg
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 11 | 12 | 12 | 12
ml/hr/kg
  Day 1 | 2459 (897) | 2285 (1103) | 2697 (1285) | 2320 (1375)
  Week 2 | 1828 (919) | 1509 (482) | 2047 (771) | 1777 (476)

16. Secondary Outcome: Pharmacokinetic (PK) Assessments t(1/2)
Description: Plasma concentrations of vamorolone were measured using a specific and validated liquid chromatography tandem mass spectrometry (LC-MS) assay. t1/2= elimination half life.
Time Frame: Day 1, Week 2
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 11 | 12 | 12 | 12
hour
  Day 1 | 2.1 (0.85) | 1.8 (0.43) | 1.9 (0.79) | 1.9 (0.95)
  Week 2 | 1.9 (0.96) | 2.1 (0.8) | 1.9 (1.02) | 1.4 (0.35)

17. Secondary Outcome: Pharmacokinetic (PK) Assessments (Cmax)
Description: as for outcome 15
Time Frame: Day 1, Week 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
Number analyzed (Participants) | 11 | 12 | 12 | 12
ng/mL
  Day 1 | 22.9 (13.4) | 75.9 (25.9) | 199 (111) | 855.6 (471)
  Week 2 | 32.2 (15.2) | 124.7 (42.5) | 252.2 (96) | 970 (270)

18. Secondary Outcome: Metabolites in Safety Testing (MIST) Assessment
Description: A portion of each blood sample of the Week 2 (Day 14) pharmacokinetic assessment time points for the subjects receiving vamorolone 2 mg/kg/day was used for analysis of vamorolone metabolites.
Time Frame: Week 2 (Day 14)
Measure: Mean (Standard Deviation); unit: % of total drug related exposure
Arm/Group | Dose Level Group 3
Number analyzed (Participants) | 12
% of total drug related exposure
  M1 | 34.42 (2.79)
  M2 | 1.16 (0.06)
  M3 | 1.21 (0.07)
  M4 | 37.84 (3.78)
  M5 | 2.73 (0.17)
  Vamorolone | 22.64 (0.69)

ADVERSE EVENTS:
Time Frame: Adverse events will be recorded from the date of informed consent and through the time of the subject's last study visit. Serious adverse events will be recorded from the date of informed consent and for up to 30 days after final drug administration.
Description: The incidence of TEAEs will be summarized by dose level, SOC and preferred term; dose level, SOC, and intensity (CTCAE grade; CTCAE version 4.03); dose level, SOC, and outcome; and dose level, SOC and relationship to study drug.
Arm/Group | Dose Level Group 1 | Dose Level Group 2 | Dose Level Group 3 | Dose Level Group 4
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 7/12 | 6/12 | 8/12 | 7/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level Group 1 (N=12) | Dose Level Group 2 (N=12) | Dose Level Group 3 (N=12) | Dose Level Group 4 (N=12)
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Faeces Discoloured (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lip Swelling (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Enterobiasis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0
Lice Infestation (Infections and infestations) | 0 | 0 | 1 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 3 | 2 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1
Emotional Disorder (Psychiatric disorders) | 0 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 1 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash Macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-01-20): https://cdn.clinicaltrials.gov/large-docs/64/NCT02760264/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/64/NCT02760264/SAP_001.pdf